CLINICAL TRIAL: NCT00009672
Title: Morphine, Nortriptyline and Their Combination in Sciatica Treatment
Brief Title: Pain Treatment for Sciatica
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 010076; 01-D-0076
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-12-12

CONDITIONS: Radiculopathy; Sciatica
Keywords: Low Back Pain; Opioid; Antidepressant; Randomized Controlled Trial; Analgesic; Sciatica
MeSH Terms: conditions — Radiculopathy; Sciatica; Low Back Pain | interventions — Nortriptyline; Morphine

INTERVENTIONS:
Drug: Nortriptyline
Drug: Morphine

SUMMARY:
This study will test the effectiveness of two drugs-nortriptyline and MS Contin (a type of morphine)-to treat pain caused by lumbar radiculopathy, or sciatica. Sciatica results from damage to the lumbar nerve roots, typically causing back pain and sharp, shooting pain down one or both legs. Although sciatica is common, there are no good treatments for it. Tricyclic antidepressants, such as nortriptyline, and opioids, such as morphine, have been effective in treating other kinds of pain from nerve damage.

Patients between 18 and 65 years of age who have had sciatica pain daily for at least 3 months may be eligible for this study.

Participants will provide a medical history and occupational and other social information. They will undergo a neurological examination, routine blood tests and an electrocardiogram and will fill out three questionnaires providing information on daily functioning and psychological well-being.

This "cross-over" study consists of several parts, including a baseline study and four different treatment regimens. During each part, patients keep a daily log in which they rate their pain, record other procedures they undergo, such as injections and manipulations, and record medication side effects.

In the first week of the study, patients remain on their current medications. Any antidepressants or opioids are stopped gradually before starting the drug trials. After the first week, patients go through the following four drug trials in random order:

1. Nortriptyline and inert placebo-Patients take nortriptyline in doses ranging from 25 mg. to 100 mg. and an inert placebo for morphine. (An inert placebo is a dummy pill; it looks like the test drug but has no active ingredient.)
2. MS Contin (morphine) and inert placebo-Patients take MS Contin in doses ranging from 30 mg. to 90 mg. and an inert placebo for nortriptyline.
3. Nortriptyline and MS Contin-Patients take MS Contin and nortriptyline in the same dose ranges as for each drug alone.
4. Active placebo and inactive placebo-Patients take an active placebo-in this case benztropine-and an inert placebo. An active placebo is a drug that does not work for the problem being studied but whose side effects are like those of the test drug-in this case, slight sleepiness or dry mouth. Benztropine is given at one-third the recommended dosage.

For each drug regimen, the medication dose is increased gradually over 5 weeks until the maximum tolerated dose is reached. At the end of each regimen, patients are taken off the study drugs over a 12-day tapering period and are off drugs completely for another 2 days.

Patients are seen by a doctor or nurse at the 7-week point in each study period. After all the drug trials are finished, patients repeat the questionnaires they filled out at the beginning of the study. Patients and their doctors will be informed of the medications that were effective in each individual's care.

DETAILED DESCRIPTION:
Irritation or damage to lumbar nerve roots referred to as lumbar radiculopathy or sciatica is a very common clinical entity with a lifetime prevalence of 1-3% in the adult population. Lumbar radiculopathy typically causes back pain and sharp, shooting pain in the leg(s). Despite its prevalence and disabling characteristics, sciatica has never been selectively studied in drug trials. It is plausible to assume that tricyclic antidepressants and opioids, which are effective in the treatment of other neuropathic pain syndromes will be beneficial for chronic lumbar radicular pain as well. This is a randomized, double-blind, placebo-controlled, four period cross-over study of chronic lumbar radicular pain. Patient selection will target men and women of all ethnic backgrounds between the ages of 18 and 65 who have had signs and symptoms of sciatica for 3 months or more. Treatments are: 1. nortriptyline (25-100 mg); 2. morphine (MS Contin 30-90 mg); 3. nortriptyline (25-100 mg) plus morphine, (MS Contin 30-90 mg); 4. combination of an active placebo, benztropine (0.25-1 mg) and an inert placebo. Patients will be called twice a week to individually titrate doses and monitor side effects. The primary outcome measures in this study will be the daily pain scores in the low back, in the leg and combined. Patients' quality of life and activities of daily living will be secondary outcome measures as assessed by the SF 36 and Oswestry and the Beck questionnaires. Fifty one patients will be enrolled in this study and the duration of the study will be 37 weeks.

ELIGIBILITY:
* INCLUSION CRITERIA:

In this study chronic lumbar radicular signs and symptoms are defined as pain located in the lower lumbar spine corresponding to L1 and below for at least 3 months with radicular characteristics, i.e. pain described as sharp, burning, with numbness and/or tingling.

Ability to understand the study measures and mentally capable of give consent to participate in the study (based on an 8th grade education level)

Willingness to refrain from taking opioids other than their study medication.

Patients with failed back syndrome who satisfy the criteria outlined in Appendix II.

Patients with a pain level of 4/10 or greater on a scale of 0 to 10.

EXCLUSION CRITERIA:

Major coexisting medical condition such as cancer, chronic obstructive pulmonary disease and severe hepatic and renal dysfunction.

Prostatic disease requiring usage of urological medications.

Pregnancy or lactation.

Unwillingness to discontinue pain medication(s) at study onset as follows: narcotic pain medications, tricyclic antidepressants (TCAs), selective serotonin reuptake inhibitors (SSRIs) and monoamine oxidase inhibitors (MAOIs).

Presence of pain of greater intensity in any other location than the low back or leg.

Current major depression requiring usage of antidepressants.

History of narcotic abuse at any time in the past and/or drug or alcohol abuse in the past year.

History of narrow angle glaucoma.

History of epilepsy.

Current symptoms of coronary artery disease.

History of fibromyalgia as described by Wolfe F et al., (1990) (a minimum of 12 out of 19 points of tenderness must be present to satisfy criteria for fibromyalgia).

History of spinal unstability (based on an MRI finding of grade II spondylolisthesis or greater).

Cognitive impairment such that the individual is unable to give informed consent, complete study data collection tools or required study visits.

Unwillingness to use adequate contraception (such as birth control pills or barrier methods with spermicide simultaneously).

Presence of other medical condition presenting with numbness and pain in lower extremities, such as diabetic polyneuropathy and peripheral vascular disease.

Allergy to any of the medications used in the study.

Age 18 years or less due to rarity of sciatica in this age group.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2001-01-30; Study Completion 2006-12-12

PRIMARY OUTCOMES:
Daily overall pain level, pain in the low back and pain in the lower extremities will be rated on a scale of 0 to 10.

SECONDARY OUTCOMES:
End of each treatment period: Pain symptoms, Use of other meds,Use of other non-meds, questionnaires, Oswestry and Beck Depression, Disability,Patients' global satisfaction with the study medications during the period.
End of Study: Patient preference.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Dellemijn P. Are opioids effective in relieving neuropathic pain? Pain. 1999 Apr;80(3):453-462. doi: 10.1016/S0304-3959(98)00256-5. PMID 10342407